CLINICAL TRIAL: NCT05570591
Title: Subthreshold Nanosecond Laser for Non-resolving Central Serous Chorioretinopathy: A Double-masked Sham-controlled Randomised Trial
Brief Title: Subthreshold Nanosecond Laser for Non-resolving Central Serous Chorioretinopathy
Acronym: NANO-C
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Eye Medical Pty Ltd. (Industry)
Collaborators: Center for Eye Research Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NANO-C
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Central Serous Chorioretinopathy
Keywords: Subthreshold nanosecond laser; Laser; 2RT; CSR; Central Serous Chorioretinopathy; Chorioretinopathy
MeSH Terms: conditions — Central Serous Chorioretinopathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active laser (Active Comparator): Application of the active 2RT sub threshold laser
  Interventions: Device: 2RT subthreshold nanosecond laser - active
- Sham laser (Sham Comparator): Application of sham laser (i.e. flashing lights which replicate the look of active laser to the participant)
  Interventions: Device: 2RT subthreshold nanosecond laser - sham

INTERVENTIONS:
Device: 2RT subthreshold nanosecond laser - active — The 2RT™ Q-switched YAG laser (532nm) delivering 3 nanosecond pulses; 400 um spot size, is a pulsed subthreshold nanosecond (SNL) laser, which uses low energy levels to produce limited effects that selectively target melanosomes within the pigmented retinal pigment epithelial (RPE) cells.
  Other Names: 2RT; SNL
  Arms: Active laser
Device: 2RT subthreshold nanosecond laser - sham — Application of sham laser (i.e. flashing lights which replicate the look of active laser to the participant) from the 2RT subthreshold nanosecond laser device.
  Other Names: Sham laser
  Arms: Sham laser

SUMMARY:
This is a prospective, multicentre, sham-controlled, participant- and assessor-masked superiority trial with two parallel treatment arms which aims to investigate the safety and efficacy of subthreshold nanosecond laser (SNL) in a series of adults with sub-retinal fluid secondary to non-resolving central serous chorioretinopathy (CSCR) by visual and anatomical outcomes.

The study population will be individuals with adults (aged 18-70 years inclusive) with non-resolving CSCR (defined as CSCR present for a duration of more than 3 months presenting with either focal or diffuse leakage) who meet all eligibility criteria.

60 subjects total will be enrolled into the study - 40 randomized to receive SNL treatment and 20 to receive sham treatment as per a 2:1 randomization schedule and stratified by type of CSCR (focal vs diffuse).

The study has a 24-week study period with five scheduled visits: screening, randomisation (first treatment), 6-week follow up (with second treatment where eligible), 12-week follow-up , 18-week follow-up, and 24-week follow-up.

The primary outcome is the proportion of laser-treated study eyes that show resolution of sub-retinal fluid (SRF) as observed on optical coherence tomography (OCT) compared to sham-treated study eyes at 24 weeks.

The safety endpoint will be proportion of laser-treated eyes that lose ≥10 letters of of vision (measured on a standard vision chart) compared to sham-treated study eyes and fellow eyes over 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years
2. Both males and females
3. Individuals with non-resolving CSCR as defined by presence of any SRF on OCT for > 3 months from date of diagnosis to randomisation visit
4. BCVA of 35 to 80 letters (Snellen equivalent of 6/6 to 6/60) in the study eye
5. Ability, willingness and sufficient cognitive awareness to consent to the trial, received randomised SNL treatment or sham procedure, and complete all visits as per the study schedule

Exclusion Criteria:

1. A need for extraneous, continuous steroids to control any disease, including both systemic steroids (e.g., for systemic autoimmune conditions) and ocular steroids (e.g., for uveitis), or ongoing anabolic steroid use
2. Any systemic disease that leads to elevated endogenous steroid levels including raised 24h urinary cortisol level > 100 ug/24h consistent with Cushing's syndrome
3. Any ocular disease in the study eye, other than CSCR, which in the opinion of the investigator may significantly compromise assessment of the retina, or which would compromise the ability to assess any effect following SNL treatment including, but not limited to:

   * Age related macular degeneration
   * Any evidence of a neovascular membrane in the macular (either exudative or non-exudative)
   * Diabetic retinopathy (unless limited to fewer than 10 microaneurysms and/or small retinal haemorrhages, without retinal thickening on OCT)
   * Macular pathology or pigmentary abnormalities including but not limited to: pattern dystrophy, myopic maculopathy, angioid streaks, resumed ocular histoplasmosis syndrome, visually-significant epiretinal membranes, macular hole or pseudohole
   * Optic nerve pathology, including optic atrophy, history of optic neuropathy
   * Myopic crescent wider than 50% of the longest diameter of the optic disc, or closer than 1500 µm to the fovea
   * Retinal vascular diseases including branch or central vein or artery occlusion
   * Choroidal nevus within 2 DD of the fovea associated with depigmentation or overlying drusen, if these drusen are used to determine eligibility
   * Active uveitis or ocular inflammation
   * Corneal pathology precluding visualization of fundus or increasing the risk of using a contact lens, such as corneal dystrophy, recurrent corneal erosion syndrome or sensitivity to the application of a contact lens
4. History or presence of uncontrolled glaucoma or raised intraocular pressure which would preclude safe dilation of the pupil to allow adequate assessment and application of SNL treatment
5. History of prior laser surgery to the retina including subthreshold laser (focal retinopexy for a peripheral retinal tear performed more than 90 days prior to the entry into the study is permitted)
6. Significant cataract or other ocular media which, in the opinion of the investigator, significantly limits the visual acuity or view of the retina
7. Cataract surgery within three months preceding baseline, or a history of post-operative complications within the last 12 months preceding baseline in the study eye (uveitis, cyclitis, etc.)
8. Previous retinal or ocular surgery, the effects of which may now or in the future complicate assessment of CSCR (routine cataract surgery more than 3 months prior is permitted)
9. Known hypersensitivity to fluorescein
10. Use of any systemic or ocular medication known to be toxic to the retina, excluding tamoxifen unless there is evidence of toxicity
11. Pregnant or lactating women
12. Current participation in any other investigational ophthalmological clinical trial
13. Other health-related reasons which make an individual inappropriate for participation in this study based on the investigator's medical judgment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Resolution of sub-retinal fluid in study eyes | 24 weeks
  The change in amount of sub-retinal fluid (SRF) as observed on optical coherence tomography (OCT) imaging in the SNL-treated compared to sham-treated study eyes over 24 weeks.

OTHER OUTCOMES:
Safety Endpoint | 24 weeks
  The proportion of eyes that lose ≥10 letters of best corrected visual acuity (BCVA) in the SNL-treated compared to sham-treated study and fellow eyes over 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Mali Okada, MBBS FRANZCO, Principal Investigator — Center for Eye Research Australia
Locations (2):
- Australia (2):
  - Centre for Eye Research Australia, East Melbourne, Victoria
  - Retinology Institute, Glen Iris, Victoria

IPD SHARING:
Plan to Share IPD: No